CLINICAL TRIAL: NCT06259162
Title: The Evaluation the Relationship Between LAG-3 Expression / Immune Checkpoint Protein Expression and Neoadjuvant Chemotherapy Plus Immune Checkpoint Inhibitor in Triple Negative Breast Cancer
Brief Title: LAG3 Expression in Triple Negative Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, JI-YEON, KIM, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: LAG3_Breast
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Triple Negative Breast Cancer; Immune Checkpoint Inhibitor
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LAG-3 expression/immune checkpoint protein expression evaluation (Experimental)
  Interventions: Procedure: LAG-3 expression / immune checkpoint protein expression

INTERVENTIONS:
Procedure: LAG-3 expression / immune checkpoint protein expression — Evaluate the tissue and blood before and after chemotherapy

SUMMARY:
This study is the experimental study for relationship between LAG-3 expression / immue checkpoint protein expression and neoadjuvant chemotherapy plus immune checkpoint inhibitor in triple negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Planned neoadjuvant chemotherapy
* Triple negative breast cancer

Exclusion Criteria:

* HER2-positive breast cancer
* Hormone receptor positive breast cancer

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
LAG-3 expression/immune checkpoint preotein expression | Before chemotherapy, 1 weeks & 3 weeks after chemotherapy, curative surgery
  Relationship neoadjuvant chemotherapy plus immune checkpoint inhibitor

CONTACTS AND LOCATIONS:
Locations (1):
- Ji-Yeon Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No